CLINICAL TRIAL: NCT03186261
Title: Evaluation of the Antibacterial Effect of Nano Silver Fluoride Versus Chlorhexidine on Occlusal Carious Molars Treated With Partial Caries Removal Technique: A Randomized Clinical Trial
Brief Title: Antibacterial Effect of Nano Silver Fluoride vs Chlorhexidine on Occlusal Carious Molars Treated With Partial Caries Removal Technique
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, ali mostafa shamaa, Principle Investigator, Dentist at Suez health directorate, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: amshamaa
Record Dates: First submitted 2017-06-10; First posted 2017-06-14 (Actual); Results first posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-08

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries | interventions — Bisco Cavity Cleanser; chlorhexidine gluconate; Solutions

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Nano silver fluoride solution (Experimental): Nano silver fluoride solution (Prepared in Nanotech Co., Egypt) based on silver nanoparticles, chitosan and fluoride. Each tooth will receive two drops of NSF with a micro brush, equivalent to a dose of 10 mg of the solution.
  Interventions: Drug: Nano silver fluoride solution
- Cavity Cleanser (Active Comparator): Chlorhexidine digluconate 2 % solution (Cavity Cleanser, Bisco, USA). Each tooth will receive two drops of cavity cleanser with a micro brush, equivalent to a dose of 10 mg of the solution.
  Interventions: Drug: Cavity Cleanser

INTERVENTIONS:
Drug: Nano silver fluoride solution — Nano silver fluoride that composed of silver nanoparticles, chitosan and fluoride that combines preventive and antimicrobial properties.
  Other Names: NSF
  Arms: Nano silver fluoride solution
Drug: Cavity Cleanser — Moistens dentin surface after cavity preparation using a micro brush.
  Other Names: Chlorhexidine digluconate 2 % solution
  Arms: Cavity Cleanser

SUMMARY:
* The teeth of the patients that meet inclusion criteria will be anesthetized, isolated with a rubber dam.
* Cavity opened using conventional high-speed rotary instruments.
* The central cariogenic biomass and the superficial parts of the necrotic dentine will be removed with round burs.
* Caries lesion will be completely removed in the enamel/dentin junction.
* The excavation procedure will be terminated as soon as the soft and wet dentine was removed and the remaining tissue was leathery but not hard on exploring.
* A dentinal sample will then be collected from the base of the cavity using sterile spoon excavator as a baseline for bacteriological assessment.
* Then, application of either intervention or control agent, another dentinal sample will be collected using a sterile excavator and transferred into sterile tubes and transferred to the laboratory for microbiological analysis.
* Filling of the cavity with resin composite restoration.
* All clinical procedures will be carried out at the same visit.

DETAILED DESCRIPTION:
I.1. Study setting This clinical study will be held in the Clinic of Conservative Dentistry Department, Faculty of Dentistry, Cairo University, Egypt. The researcher will bear ultimate responsibility for all activities associated with the conduct of a research project including recruitment of patients, explaining and performing the procedures to them.

II.4.a Excavation protocol:

The teeth of the patients that meet inclusion criteria will be anesthetized, isolated with a rubber dam. Cavity opened using conventional high-speed rotary instruments. The central cariogenic biomass and the superficial parts of the necrotic dentine will be removed with round burs. Caries lesion will be completely removed in the enamel/dentin junction. The excavation procedure will be terminated as soon as the soft and wet dentine was removed and the remaining tissue was leathery but not hard on exploring. A dentinal sample will then be collected from the base of the cavity using sterile spoon excavator as a baseline for bacteriological assessment. Then, application of either intervention or control agent, another dentinal sample will be collected using a sterile excavator and transferred into sterile tubes and transferred to the laboratory for microbiological analysis.

II.4.b Assessment of Outcome:

Samples of carious dentine will be collected with sterile excavator before and after application of intervention/control agent. The dentine samples will be transferred to sterile container containing a 1mL thioglycollate medium used as a carrier, then this sterile container will be kept in an ice box and taken to the microbiology laboratory for processing, within an hour, by another examiner who is blinded to the type of agent applied after partial caries removal. Samples will be vortexed for two minutes, decimally diluted and 0.1 ml will be plated on Mitis Salivarius Bacitracin agar plates, these plates will be incubated anaerobically for 48 hour at 37ºC then aerobically for 24 hour at room temperature. The number of colonies will be expressed as colony-forming units (CFU/ml) compared before and after application of the antibacterial agent.

II.5. Participant timeline:

All clinical procedures will be carried out at the same visit.

II.6. Sample size calculation:

The aim of this study is to evaluate the antibacterial action Nano Silver Fluoride solution application in comparison to Chlorhexidine solution after partial caries removal in class I carious permanent molar. Based on a previous study by Mohan et al. 20165, the expected difference between two interventions is expected to be 2.1±2.2CFU/mL × 103. Using power 80% and 5% significance level we will need to study 18 in each group to be able to reject the null hypothesis that the population means of the experimental and control groups are equal. This number is to be increased to 22 patients in each group to compensate for possible losses during follow up. The sample size was calculated by PS program.

II.7. Recruitment:

Patients will be recruited from outpatient clinic of Conservative Dentistry Department in Faculty of Dentistry, Cairo University; after explaining the benefits/risks from the application of the interventions, then eligible patients will be recruited to fulfil the eligibility criteria according to participant timeline.

II.8.a. Recruitment Strategy:

The patients will be subjected to full examination and diagnosis using dental charts. Once the patients that are potentially eligible for this study are identified, they will be contacted by the researcher who will explain the study and ascertains the patient's interest. If interested, more detailed evaluations and preparations are made.

II.9. Randomization and assignment of interventions:

II.9.a. Allocation sequence generation:

The allocation sequence will be generated using (www.randomization.com).

II.9.b. Allocation concealment mechanism:

The randomization unit was the tooth, and the randomization procedure will be performed as follows. A number corresponding to each treatment group will be printed on pieces of paper and kept in dark containers. A paper will be selected from the container by a person other than the operator, and the treatment indicated will be performed (intervention/control). Blinding of the operator is not possible, because the color of intervention and control solution is different. The operator is blinded until randomization into groups, to avoid biases with regard to the application of antibacterial agent. Also, the examiner who will carry the microbiological analysis of dentin samples will be blinded to the type of agent applied during treatment. Finally, the treatment results will be assessed blindly by a statistician.

II.9.c. Implementation:

Dr. Mai Mamdouh (co-supervisor) will perform the allocation sequence and assign the participants to the intervention/Control treatment group.

II.9.d. Blinding:

The side to which interventions or control is assigned to will be recorded and all records of all patients will be kept with the main supervisor. Blinding of the operator is not possible, because the color of intervention and control solution is different. The operator is blinded until randomization into groups, to avoid biases with regard to the application of antibacterial agent. Also, the examiner who will carry the microbiological analysis of dentin samples will be blinded to the type of agent applied during treatment. Finally, the treatment results will be assessed blindly by a statistician.

II.10. Data collection methods:

*Baseline data collection: For every patient medical history, dental history and examination charts will be filled by the operator. The report will be anonymous where patients identified by their serial numbers (the first letter of the first and last name and date of birth) only will be registered. Full detailed personal data of the patient will be written in separate sheet having the patient's serial number for further contact with patient.

*Outcome data collection: The results will be converted into a table to facilitate the description of the results. The microbiological analysis will be performed blindly in relation to the type of solution applied after partial caries removal.

II.11.Data management:

The data will be entered and stored on a personal computer. Double data entry will be saved on an external hard disc to prevent loss of data.

II.12. Statistical methods:

Data will be analyzed using IBM SPSS advanced statistics (Statistical Package for Social Sciences), version 21 (SPSS Inc., Chicago, IL). Numerical data will be described as mean and standard deviation or median and range. Categorical data will be explored for normality using Kolmogrov-Smirnov test and Shapiro-Wilk test. Comparisons between two groups for normally distributed numeric variables will be done using the Student's t-test while for non normally distributed numeric variables will be done by Mann-Whitney test. Comparisons between categorical variables will be performed using the chi square test. A p-value less than or equal to 0.05 will be considered statistically significant. All tests will be two tailed.

II.13. Monitoring:

II.13.a. Data monitoring:

The main supervisor will monitor this study. His role is to monitor any risk of bias could be done from participants, operator or assessors. Also to monitor blinding of the assessors and patient safety, outstanding benefits or harms.

II.13.b. Harms:

The main supervisor should inform participants about the possible harms, if present. Participants are allowed to contact the operator at moment through telephone. In case of accidental pulp exposure during excavation , emergency access cavity and pulp extirpation will be done by the operator and then the patient will be referred to Endodontic Department clinic to complete the rool canal treatment.

II.13.c. Auditing:

In the present trial, auditing will be done by the main and co-supervisors to assure quality of the research frequency procedures.

II.14. Ethics and dissemination

II.14.a. Research ethics approval:

Application forms for carrying out the clinical trial, checklist and informed consent of Research Ethics Committee (REC) Faculty of Dentistry, Cairo University will be retrieved and filled, then will be delivered for (REC) committee for approval. This is done to prevent any ethical problems during the study or any harm for any of the participants.

II.14.b. Protocol amendments:

If a new protocol will be used a protocol amendment will be submitted; containing a new copy of the new protocol and brief explanation about the differences between it and the previous protocols. If there is a change in the existing protocol that affects safety of subjects, investigation scope or scientific quality of the trial, an amendment containing a brief explanation about the change will be submitted. If a new author will be added to accomplish the study, an amendment including the investigator's data and qualifications to conduct the investigation will be submitted to prevent ghost authorship.

II.14.c. Consent:

The operator (Ali Mostafa Shamaa) is responsible for admitting and signing the written consents during the enrolment day.

II.15. Confidentiality:

Name, personal data and pictures of the participants will not appear on the protocol form and will be maintained secured for 10 years after the trial. This is done for protection of participants' privacy and civil rights.

II.16. Declaration of interests:

There is no conflict of interest, no funding or material supplying from any parties.

Access to final data will be allowed to the operator ,the main and co-supervisors of the study who are not involved in assessment of the outcome.

II.18. Ancillary and post-trial care:

Patients will be followed up after the application after 3, 6 months.

II.19. Dissemination policy:

Full protocol will be published online in www.clinicaltrials.gov to avoid repetition and to keep the integrity of the research work. Thesis will be discussed in front of judgment committee. The study will be published to report the results of this clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria of participants:

  1. Not received antibiotic therapy since 1 month before sampling.
  2. Good oral hygiene.
  3. Co-operative patients approving the trial.
* Inclusion Criteria of teeth:

  1. Class I deep caries lesions in permanent molar (reaching ≥ 1/2 of the dentin on radiographic examination).
  2. Absence of spontaneous pain; negative sensitivity to percussion; and absence of periapical lesions (radiographic examination).

Exclusion Criteria:

* Exclusion criteria of participants:

  1. Pregnancy.
  2. Systemic disease or severe medical complications.
  3. Heavy smoking.
  4. Xerostomia.
  5. Lack of compliance.
* Exclusion criteria of teeth:

  1. Class II caries lesion.
  2. Shallow or enamel caries.
  3. Cuspal loss or caries beneath the gingival margin.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randa Hafez, PHD, Study Director — Cairo University; Mai Mamdouh, PHD, Study Chair — Cairo University
Locations (1):
- Faculty of Dentistry, Cairo University., Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Mohan PV, Uloopi KS, Vinay C, Rao RC. In vivo comparison of cavity disinfection efficacy with APF gel, Propolis, Diode Laser, and 2% chlorhexidine in primary teeth. Contemp Clin Dent. 2016 Jan-Mar;7(1):45-50. doi: 10.4103/0976-237X.177110. PMID 27041900

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Teeth
Period: Overall Study
Arm/Group | Nano Silver Fluoride Solution | Cavity Cleanser
Started | 22; 22 Teeth | 22; 22 Teeth
Completed | 22; 22 Teeth | 22; 22 Teeth
Not Completed | 0; 0 Teeth | 0; 0 Teeth

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nano Silver Fluoride Solution | Cavity Cleanser | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 22 | 44
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 14 | 30
  Male | 6 | 8 | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Egypt | 22 | 22 | 44
Vital Permanent molar with deep occlusal carious lesion [Number; unit: Teeth] | 22 | 22 | 44

OUTCOME MEASURES:

1. Primary Outcome: Bacterial Count of Streptococus Mutans
Description: Digital Colony Counter, Agar Diffusion test
Time Frame: 5 minutes on average between baseline and after application of the solution
Measure: Mean (Standard Deviation); unit: CFU/ml log10
Arm/Group | Nano Silver Fluoride Solution | Cavity Cleanser
Number analyzed (Participants) | 22 | 22
CFU/ml log10
  Baseline | 2.00 (0.33) | 2.04 (0.23)
  After solution application | 1.12 (0.59) | 1.05 (0.63)

ADVERSE EVENTS:
Time Frame: 6 month
Arm/Group | Nano Silver Fluoride Solution | Cavity Cleanser
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-03-02): https://cdn.clinicaltrials.gov/large-docs/61/NCT03186261/Prot_SAP_ICF_000.pdf